CLINICAL TRIAL: NCT06455644
Title: The Accuracy of Left Atrial Appendage Occluder Size Selection Between Preoperative CT and Intraoperative DSA Evaluation During a Combined Atrial Fibrillation Ablation and Left Atrial Appendage Occlusion Procedure
Brief Title: Accuracy of LAA Occluder Size Selection: CT vs. DSA During Combined AF Ablation and LAA Occlusion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Shantou University Medical College (Other)
Responsible Party: Principal Investigator, Zhongbo Xiao, Chief physician, First Affiliated Hospital of Shantou University Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-2024-091
Record Dates: First submitted 2024-06-04; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Atrial Fibrillation; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases
Keywords: Left atrial appendage closure; Atrial fibrillation; Pacifier-like occluder; Stroke prevention
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT group (Experimental): CT-Guided Size Selection for LAA Occluder
  Interventions: Other: CT group
- DSA group (Active Comparator): DSA-Guided Size Selection for LAA Occluder
  Interventions: Other: DSA group

INTERVENTIONS:
Other: CT group — After completing the AF ablation, select the appropriate LAA occluder based on preoperative CT measurements for implantation.
  Arms: CT group
Other: DSA group — After completing the AF ablation, select the appropriate LAA occluder based on intraoperative DSA measurements for implantation.
  Arms: DSA group

SUMMARY:
This study is a prospective, multi-center, randomized controlled trial. The subjects are patients scheduled to undergo a combined procedure of atrial fibrillation (AF) ablation and left atrial appendage (LAA) occlusion. After signing the informed consent form, the subjects will be randomly assigned to either the cardiac Computed Tomography (CT) group or the Digital Subtraction Angiography (DSA) group. The operator will select the appropriate LAA occluder size for implantation based on different measurement methods. All subjects will undergo clinical follow-up before discharge and at 3 months postoperatively, as well as telephone follow-up 1-5 years after the surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Patients with non-valvular atrial fibrillation scheduled to undergo atrial fibrillation ablation and percutaneous left atrial appendage occlusion;
3. Able to understand the purpose of the trial, willing to participate in the study, and the subject or their legal representative has signed the informed consent form, and is willing to complete the follow-up according to the protocol requirements.

Exclusion Criteria:

1. Allergy to contrast agents or other conditions that preclude cardiac CT or DSA imaging;
2. Absence of clear images for measuring the diameter of the LAA in all layers of the CT scan;
3. Imaging indicates the presence of thrombus in the left atrium or LAA;
4. Patients with valvular AF (mechanical valve replacement or moderate to severe mitral stenosis combined with AF);
5. LAA depth < 15 mm, or LAA anchor zone diameter < 10 mm or > 33 mm;
6. Female patients of childbearing age planning to become pregnant during the follow-up period required by this study;
7. Currently participating in another clinical trial of drugs or medical devices and has not yet completed the primary endpoints of that study, which may confound the results of this study or affect the participant's compliance with the follow-up;
8. Other conditions that the investigator deems make the participant unsuitable for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Accuracy of LAA occluder size selection | During procedure
  Accuracy is defined as: the occluder's anchor disc seats beyond the circumflex artery, the compression of the anchor disc after release is 3-6 mm, peri-device leak is ≤ 3 mm, and the occluder remains stable during the tug test.

SECONDARY OUTCOMES:
Procedure success | During procedure
  Technical success of the LAA occlusion procedure without serious procedure-related complications
Peri-device leak at 3 months post-procedure | 3 months
  Proportion of peri-device leak at the occluder evaluated by TEE or CT
Procedure-related times | During procedure
  Total procedure time, AF ablation time, and LAA occlusion time
Incidence of major adverse events (MAE) related to the device or procedure within 3 months post-procedure | 3 months
  MAE is defined as unexplained death or any device or procedure-related complications, including but not limited to death, stroke, or transient ischemic attack (TIA), serious pericardial effusion/pericardial tamponade requiring pericardiocentesis or surgery, device embolization, life-threatening or severe bleeding events, and severe vascular access complications

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Foshan Nanhai District People's Hospital, Foshan, Guangdong
  - The Second People's Hospital of Foshan, Foshan, Guangdong
  - Meizhou Hospital of Traditional Chinese Medicine, Meizhou, Guangdong
  - First Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Guangdong Provincial Zhongshan Hospital of Traditional Chinese Medicine, Zhongshan, Guangdong